CLINICAL TRIAL: NCT02934165
Title: Safety Skills Training For Parents of Preschool Children
Acronym: Preschool_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBIR72RR-2; R44HD047068 (NIH)
Record Dates: First submitted 2014-12-30; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Behavior
Keywords: child safety; injury; computer; prevention; internet
MeSH Terms: conditions — Behavior; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Safety 123 (Experimental): Parents viewed a website with videos on child injury prevention strategies and received emails for 30 days inviting them to view additional videos.
  Interventions: Behavioral: Family Safety 123
- AAP TIPP sheets (Active Comparator): Parents viewed online injury prevention materials developed by the American Academy of Pediatrics and had continuing access to these materials for 30 days.
  Interventions: Behavioral: AAP TIPP sheets

INTERVENTIONS:
Behavioral: Family Safety 123 — Theoretically-based injury prevention videos for families
  Other Names: Family Safety 123 for Parents of Children 2-5
  Arms: Family Safety 123
Behavioral: AAP TIPP sheets — American Academy of Pediatrics The Injury Prevent Program materials converted to web-based materials.
  Arms: AAP TIPP sheets

SUMMARY:
As the leading cause of death and disability in children in America, unintentional injuries are a critical public health issue. Most injuries can be prevented by parents implementing effective child safety practices. This project produced an interactive multimedia (IMM) program delivered via Internet/Intranet that taught injury prevention skills to parents of children aged 2 through 5 years, with the ultimate goal of reducing mortality and disability from unintentional injury in this population.

DETAILED DESCRIPTION:
This project produced a comprehensive, interactive multimedia (IMM) program called Family Safety 123 to teach childhood injury prevention skills to parents of children 2 to 5 years of age. The program contained 40 high-quality video clips, each 2 to 5 minutes in length, depicting injury prevention strategies in 13 content areas: supervision, preventing airway obstructions, poison awareness, preventing burns, preventing falls, firearm safety, motor vehicle safety, pedestrian awareness, sports, playgrounds, water safety, bike safety, and other safety concerns. Each content area contained 1 to 6 videos comprised of short video presentations, modeling vignettes demonstrating desired behaviors, supportive testimonials, and suggestions for modifications to home and recreational environments. Family Safety 123 video content is derived from The Injury Prevention Program (TIPP) sheets developed by the American Academy of Pediatrics, which recognizes injury prevention as a primary topic for parents.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 2-5 potentially were as young as 18 years old. Parents or legal guardians could potentially be as old as 65 or older.

Exclusion Criteria:

* Only English-speaking participants were accepted because the program was developed only for English speakers. All English-speaking parents of children aged 2-5 years old who wished to participate were included. Online Survey: parents under 18 years of age were excluded because we were unable to obtain parental consent online.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Behavioral measure: Change from baseline in identification of correct/incorrect child car safety seat and booster seat situations and bicycle helmet placement situations. | 30 days and 60 days
  Parents viewed child car seat and booster seat situations and were asked whether 9 car safety seat and 7 booster seat items were correct or incorrect. Parents also viewed 2 bicycle helmet situations and were asked to identify if these were correct or incorrect.

SECONDARY OUTCOMES:
Change in knowledge of injury prevention strategies | 30 days and 60 days
  An injury prevention knowledge scale was created across all content areas. The injury prevention knowledge scale contained 41 items (e.g., "The best way to lessen the possibility of a young child choking …") for parents of younger children and 44-items for parents of older children. The injury prevention knowledge scale represents the percent of items correctly endorsed.
Change in attitudes and beliefs about injury prevention strategies | 30 days and 60 days
  An injury prevention attitudes & beliefs scale was created across all content areas (e.g., "It is never ok to use a second hand car seat even if you know the car seat has never been involved in a crash."). Thirty-four items assessed attitudes & beliefs for parents of younger children and 33-items for parents of older children (alpha = .85 for both younger and older children). All items were assessed using a 5-point Likert scale with 1 = strongly disagree to 5 = strongly agree.
Change in self-efficacy for engaging in injury prevention strategies | 30 days and 60 days
  An injury prevention self-efficacy scale was created from 36 items across all content areas for the parents of younger children and 35 items for parents of older (e.g., "I am confident that I know the safest way to store guns and ammunition") (alpha = .77 for younger children and .89 for older children.) All items were assessed using a 5-point Likert scale with 1 = strongly disagree to 5 = strongly agree.
Change in car safety knowledge of injury prevention | 30 days and 60 days
  Three items were used to assess knowledge of car safety injury prevention (e.g., "Your child should use a forward-facing safety seat until…") with the response coded as either 0 = incorrect or 1 = correct.
Change in car safety attitudes & beliefs of injury prevention | 30 days and 60 days
  Two items were used to assess attitudes and beliefs towards car safety injury prevention (e.g., "It is never ok to use a second car seat even if you know the car seat has never been involved in a crash"). Both items were assessed with a 5-point Likert scale with 1 = strongly disagree and 5 = strongly agree. Both of the attitudes & beliefs items for the car safety attitudes content area were discarded because the wording proved confusing to participants.
Change in car safety self-efficacy in performing injury prevention skills | 30 days and 60 days
  Four items were used to assess self-efficacy in performing car safety injury prevention skills (e.g., "How confident are you that you know when to transition your child into a booster seat?"). Items were assessed with a 5-point Likert scale with 1 = not at all confident and 5 = extremely confident.
Change in wheeled sports knowledge of injury prevention | 30 days and 60 days
  Two items were used to assess knowledge of wheeled sports injury prevention (e.g., "A child carrier bike seat should…") with the response coded as either 0 = incorrect or 1 = correct.
Change in wheeled sports attitudes & beliefs of injury prevention | 30 days and 60 days
  Four items were used to assess attitudes & beliefs towards wheeled sports safety injury prevention (e.g., "It is extremely important for my child to wear a helmet whenever riding his or her bike"). Items were assessed with a 5-point Likert scale with 1 = strongly disagree and 5 = strongly agree.
Change in wheeled sports self-efficacy in performing injury prevention skills | 30 days and 60 days
  Three items were used to assess self-efficacy in performing wheeled sports injury prevention skills (e.g., "How confident are you that you know how to correctly check the fit of your child's helmet?"). Items were assessed with a 5-point Likert scale with 1 = not at all confident and 5 = extremely confident.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Grilley Swartz, MPH, CHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No